CLINICAL TRIAL: NCT03041233
Title: ABLATOR Brazil - Ablation Observational Study (Registry)
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10192
Record Dates: First submitted 2017-01-24; First posted 2017-02-02 (Estimated); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Observation; Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation / Data Collection — The following data will be reviewed / collected:
  Baseline Visit: Patient demographics; Atrial fibrillation History; Cardiovascular history; Cardiac medical history.
  Ablation Procedure: Devices used; Ablation parameters; Ablation success definition and result; Operator feedback (Device combination chosen, device maneuverability, ease of use in combination with other device); Number, experience and type of attending personnel; Definition of standard of care (follow-up procedures and occurrence).
  6- and 12-month follow-up (+/- 30 DAYS): Recurrence of atrial arrhythmias: list of atrial arrhythmias since last visit, classify episodes, duration of the episodes; Changes in therapy; In case of Repeat Ablation Procedures, reconnections and new ablations will be recorded.

SUMMARY:
The purpose of this registry is to assess the performance and clinical effectiveness of a combination of St. Jude Medical (SJM)/Abbott mapping and ablation products in the treatment of subjects with atrial fibrillation (AF).

DETAILED DESCRIPTION:
The objectives of this registry are the following:

* To confirm patient safety as part of the post market surveillance study.
* To assess performance of a combination of SJM products during procedures.
* To assess the learning curve with a combination of SJM products.
* To collect operator feedback on a combination of SJM products.

All patients from participating sites who are indicated for an atrial fibrillation ablation procedure and willing to provide written Informed Consent may be enrolled in this registry.

In order to ensure a minimum level of uniformity across site practices and to enable comparison of acute and long-term effectiveness as well as procedure efficiency according to technique used, a combination of 2 types of devices from the pre-specified list must be used to be eligible in this registry.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are indicated for an atrial fibrillation ablation procedure.

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are indicated for an atrial fibrillation ablation procedure, except for pregnant women.
Sampling Method: Non-Probability Sample
Enrollment: 833 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: André Luiz D'Avila, Principal Investigator — SOS Cardio
Locations (12):
- Brazil (12):
  - Cardioritmo Eletrofisiologia e Marpasso, Fortaleza, Ceará
  - Hospital Santa Rita, Vitória, Espírito Santo
  - Vitoria Apart Hotel, Vitória, Espírito Santo
  - Santa Casa de Misericórdia da Bahia, Salvador, Estado de Bahia
  - HOME - Hospital Ortopédico e Medicina Especializada LTDA., Brasília, Federal District
  - Procardiaco, Rio de Janeiro, Rio de Janeiro
  - Unimed de Volta Redonda, Volta Redonda, Rio de Janeiro
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - SOS Cardio, Florianópolis, Santa Catarina
  - Insitituto de Moléstias Cardiovasculares - IMC, São José Do Rio Prêto, São Paulo
  - BP, São Paulo, São Paulo
  - SEMAP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled: Patients who have indication for ablation of atrial fibrillation and who were willing to provide a written consent form, except pregnant women, were included in this registry. Patients were considered enrolled in this registry at the time they signed the written consent form.
Period: Overall Study
Arm/Group | Enrolled
Started | 833
Procedure | 829
6-month Follow-up | 803
12-month Follow-up | 705
Completed | 801
Not Completed | 32
Not completed — Death | 5
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 16
Not completed — Inclusion/Exclusion Criteria Not Met | 7
Not completed — Sponsor Request | 1
Not completed — Duplicate subject | 1
Not completed — Re-ablation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enrolled
Number analyzed (Participants) | 833
Age, Customized [Count of Participants; unit: Participants]
  <29 years | 16
  30-39 years | 61
  40-49 years | 97
  50-59 years | 220
  60-69 years | 279
  70-79 years | 145
  >80 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228
  Male | 605
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Unsuccessful Treatment Rate
Description: Percent of subjects with a repeat procedure
Time Frame: up to 6 and 12 months after ablation procedure
Population: The analysis population is subjects who received atrial fibrillation (AF) ablation for which 6-month and 12-month follow-up data was available for, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 803
Participants
  6 months | 22
  12 months: number analyzed (Participants) | 705
  12 months | 21

2. Secondary Outcome: Cardiovascular Serious Adverse Event (SAE)
Description: Percent of subjects with Cardiovascular SAE.
Time Frame: up to 6 and 12 months after ablation procedure
Population: The analysis population is subjects who received AF ablation for which 6-month and 12-month follow-up data was available for, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 803
Participants
  6 months | 2
  12 months: number analyzed (Participants) | 705
  12 months | 2

3. Secondary Outcome: Death in Subjects Who Underwent an Ablation Procedure
Description: Percent of subjects experiencing death within 12 months of ablation procedure
Time Frame: up to 12 months after ablation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 829
Participants
  Death <30 days post-procedure | 3
  Death >30 days post-procedure | 2

ADVERSE EVENTS:
Time Frame: Through 12 months
Description: An adverse event was considered when it was of cardiovascular origin with potential for the following outcomes:
  * Death;
  * A serious deterioration of the patient's health, which may result in: life-threatening disease/condition; permanent incapacity of a body structure/function; prolonged hospitalization; medical/surgical intervention to prevent life-threatening illness/injury; malignant tumor; planned hospitalization for a pre-existing condition was not considered a serious adverse event.
Arm/Group | Enrolled
All-Cause Mortality (participants affected / at risk) | 5/833
Serious Adverse Events (participants affected / at risk) | 30/833
Other Adverse Events (participants affected / at risk) | 1/833
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled (N=833)
Hematoma (Injury, poisoning and procedural complications) | 5 (5)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hematoma (Vascular disorders) | 1 (1)
Drowning (General disorders) | 1 (1)
Catheter Deformation (Injury, poisoning and procedural complications) | 1 (1)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 5 (5)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death (Hepatobiliary disorders) | 1 (1)
Hematuria (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary congestion (Injury, poisoning and procedural complications) | 4 (4)
Chest Pain (Injury, poisoning and procedural complications) | 1 (1)
Skin lesion (Infections and infestations) | 1 (1)
Pericardial Effusion (Injury, poisoning and procedural complications) | 1 (1)
Bruise (Injury, poisoning and procedural complications) | 1 (1)
Car accident (General disorders) | 1 (1)
Tamponade (Injury, poisoning and procedural complications) | 1 (1)
Perioperative infarction (Injury, poisoning and procedural complications) | 1 (1)
Sinus dysfunction/asystole after interruption of flutter (Injury, poisoning and procedural complications) | 1 (1)
Muscle abscess (Infections and infestations) | 1 (1)
Hemorrhagic stroke (Nervous system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Prolonged Hospitalization (Gastrointestinal disorders) | 1 (1)
Prolonged hospitalization (Cardiac disorders) | 1 (1)
Change in medical strategy (Cardiac disorders) | 1 (1)
Suspected bacterial endocarditis (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled (N=833)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03041233/Prot_SAP_000.pdf